CLINICAL TRIAL: NCT01816880
Title: Wellderly Immune Antibodies Study, a Sub-Study of Healthy Elderly Active Longevity (HEAL) Cohort (HSC# 004789)
Brief Title: Wellderly Immune Antibodies Study, a Sub-Study of Healthy Elderly Active Longevity (HEAL) Cohort
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Wellderly Immune Antibodies
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Antibodies Involved in Healthy Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample of approximately 20mL
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Elderly: Age 90 and over Gender: Male and Female Enrolled in the Healthy Elderly (HEAL) study prior to enrollment in this sub-study Blood sample of approximately 20mL is drawn.

SUMMARY:
The aim of this sub-study is to determine whether healthy individuals over 90 years of age possess immune cells that are involved in protection from chronic disease. The immune system is well known to produce anti-cancer and other immune cells, called antibodies that can be beneficial to our health. In this study the investigators will evaluate the immune status of the healthy individuals over 90 years of age. The investigators will be focused on studying molecules known to be involved in cholesterol, cancer like those for prostate cancer and breast cancer, inflammatory diseases, and infectious diseases like influenza.

DETAILED DESCRIPTION:
The aim of this sub-study is to determine whether the Wellderly posess neutralizing antibodies targeting antigens involved in chronic disease. The humoral immune system is well known to produce anti-cancer and other antibodies that can be long lived in vivo. In this study we will evaluate the antibody status of the Wellderly with respect to neutralizing (i) molecules known to induce cholesterol like PCSK9, (ii) antibodies against cancer antigens like PMSA (prostate cancer) or Her2 (Breast cancer), (iii) antibodies against inflammatory molecules like TNFa or IL-6, (iv) antibodies that have broad neutralizing activity against infectious diseases like influenza.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 90 and over
2. Gender: Male and Female
3. Enrolled in the Healthy Elderly (HEAL) study prior to enrollment in this sub-study
4. Eligible for Blood draw
5. Be reliable, cooperative and willing to comply with all protocol-specified procedures.
6. Able to understand and grant informed consent
7. Be healthy or have mild medical conditions that may be associated with the normal aging process, including:

   * Hypertension, well controlled with no more than 3 medications
   * Osteoporosis or Osteopenia
   * Osteoarthritis
   * Benign Prostatic Hypertrophy
   * Cataracts, Glaucoma or Macular Degeneration
   * Dyslipidemia
   * Hypothyroidism
   * Pre-Diabetes/Impaired Fasting Glucose (fasting blood glucose 100-126 mg/dL, if known)
   * Basal or Squamous Cell Carcinoma

Individuals will be excluded if ANY of the following conditions apply:

EXCLUSION CRITERIA

1. Less than 90 years of age
2. Currently undergoing treatment with any investigational agents or devices within 30 preceding enrollment in this study.
3. Self-reported history or current diagnosis of significant chronic conditions including:

   * Any Cancer (including polycythemia; excluding basal or squamous cell carcinoma
   * Coronary Artery Disease, Myocardial Infarction
   * Stroke or Transient Ischemic Attack (TIA)
   * Deep Vein Thrombosis or Pulmonary Embolism
   * Chronic Renal Disease or Hemodialysis
   * Significant Auto-Immune or Inflammatory conditions such as Rheumatoid Arthritis, Lupus, Crohn's Disease, etc.
   * Alzheimer's or Parkinson's Disease
   * Diabetes (Hemoglobin A1C > 6.5% or fasting glucose > 126 mg/dL or is treated with insulin or oral diabetic medication
   * Aortic or Cerebral Aneurysm
4. Currently taking any of the following medications on a regular basis:

   * Chemotherapeutic agents (ex. Tamoxifen, Doxorubicin, Mitoxantrone, bleomycin
   * Anti-platelet or anticoagulant agents, not including Aspirin (ex. Clopidogrel/Plavix, Dipyridamole/Aggrenox/Persantine, Ticlopidine/Ticlid, Warfarin/Coumadin, Prasugrel, etc.)
   * Cholinesterase inhibitor for Alzheimer's disease (ex. Donzepril/Aricept)
   * Insulin or oral diabetic medication
5. Individual has a significant medical condition which, in the investigator's opinion, may interfere with the individual's optimal participation in the study or would potentially confound interpretation of the individual's phenotype.

Min Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Age 90 and over Gender: Male and Female Enrolled in the Healthy Elderly (HEAL) study prior to enrollment in this sub-study
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Antibodies targeting antigens involved in chronic disease | up to 2 years
  We have made phage display libraries from the antibody genes derived from Wellderly B-cells. Remarkably, we could identify specific antibodies against several targets involved in multiple chronic diseases including PCSK9, inflammatory cytokines, and influenza hemaglutinin. We hypothesize that the Wellderly may contain antibodies targeting antigens involved in chronic disease, and that these antibodies may be protective and health-promoting.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States